CLINICAL TRIAL: NCT02160977
Title: Prospective Randomized Comparative Study on the Proprioception of the Knee Post MIS TKA (Minimally Invasive Surgery Total Knee Arthroplasty) and MIS-QS(Quadriceps Sparing ) TKA
Brief Title: Proprioception of the Knee Post MIS TKA and MIS-QS TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jia-kuo yu (Other)
Responsible Party: Sponsor-Investigator, Jia-kuo yu, professor, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QS-YU
Record Dates: First submitted 2014-06-05; First posted 2014-06-11 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Osteoarthritis
Keywords: Surgical procedures; Minimally invasive; Arthroplasty; Knee
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- QS-TKA (Experimental): patients underwent minimally invasive surgery quadriceps sparing total knee arthroplasty (MIS-QS TKA)
  Interventions: Procedure: total knee arthroplasty
- MIS-TKA (Active Comparator): patients underwent minimally invasive surgery total knee arthroplasty (MIS TKA)
  Interventions: Procedure: total knee arthroplasty

INTERVENTIONS:
Procedure: total knee arthroplasty
  Other Names: total knee replacement

SUMMARY:
If the proprioception of the affected knee post total knee arthroplasty (TKA) can recover earlier, it will accelerate the regaining of motion control ability and motion control accuracy of the TKA patients. This study compared the proprioception difference of the post operation knees between the MIS-QS TKA group and the MIS TKA group.The differences of proprioception recovery were analyzed following the two different TKA procedures and the advantages of MIS-QS TKA in the recovery of knee. proprioception were discussed.

DETAILED DESCRIPTION:
Patients were scheduled prospectively to undergo total knee arthroplasties were randomly assigned to receive either a MIS-QS TKA or a MIS TKA. Proprioception of the knee position sense was assessed by the knee angle reproduction test (10~20 degree, 30~40 degree, 80~90 degree of the knee flexion) prior operation, and 1 week, 6 weeks, 3 months and 6 months post operation. Paired two-tailed t tests with a level of significance of p < 0.05 were used to assess the effect of the different arthroplasty procedure on the postoperative knee joint proprioception for all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of osteoarthritis
* Indication of TKA

Exclusion Criteria:

* Bilateral total knee replacements
* Rheumatoid arthritis
* Genu valgus over than 10 degrees and genu varum over 15 degrees
* ROM (Range of motion) of preoperative knee joint less than 100 degree.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-10; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JIa-Kuo Yu, Doctor, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From October of 2011 to June of 2012, patients who suffered from severely osteoarthritis were recruited in this study.All the patients were hospitalized patients at Peking University Third Hospital.Patients were randomly divided into two groups by digital random method.
Pre-assignment Details: Patients refused to receive MIS-QS TKA or MIS TKA.
Groups:
- MIS-TKA: patients underwent minimally invasive surgery total knee arthroplasty (MIS TKA)
  total knee arthroplasty
- QS-TKA: patients underwent minimally invasive surgery quadriceps sparing total knee arthroplasty (MIS-QS TKA)
  total knee arthroplasty
Period: One Week After Surgery
Arm/Group | MIS-TKA | QS-TKA
Started | 45 | 45
Completed | 45 | 45
Not Completed | 0 | 0
Period: Six Weeks After Surgery
Arm/Group | MIS-TKA | QS-TKA
Started | 45 | 45
Completed | 44 | 45
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Three Months After Surgery
Arm/Group | MIS-TKA | QS-TKA
Started | 44 | 45
Completed | 44 | 43
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2
Period: Six Months After Surgery
Arm/Group | MIS-TKA | QS-TKA
Started | 44 | 43
Completed | 42 | 42
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QS-TKA | MIS-TKA | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (6.1) | 64.5 (7.1) | 65.4 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 32 | 68
  Male | 6 | 10 | 16
Preoperative HSS score,Continuous [Mean (Standard Deviation); unit: units on a scale] — Scale Name:score scale range:0~100,and a higher values represent a better outcome
  units on a scale | 56.2 (13.8) | 59.9 (14.6) | 58.1 (14.3)

OUTCOME MEASURES:

1. Primary Outcome: Proprioception of the Knee Post Operation
Description: Proprioception of the knee position sense was assessed by the knee angle reproduction test (10~20 degree, 30~40 degree, 80~90 degree of the knee flexion) prior operation, and 1 week, 6 weeks, 3 months and 6 months post operation.
  Scale Name:degree scale range:0~180 degree,and a higher values represent a worse outcome
Time Frame: six months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MIS-TKA | QS-TKA
Number analyzed (Participants) | 42 | 42
units on a scale
  preoperative proprioception at 10 ~ 20 degree | 10.3 (6.8) | 6.3 (2.9)
  preoperative proprioception at 30 ~ 40 degree | 7.3 (3.2) | 6.4 (2.1)
  preoperative proprioception at 80 ~ 90 degree | 8.0 (3.2) | 7.0 (3.7)
  one week after operation at 10 ~ 20 degree | 8.6 (2.8) | 5.0 (1.3)
  one week after operation at 30 ~40 degree | 6.3 (1.9) | 4.0 (1.5)
  six weeks after operation at 10 ~ 20 degree | 7.7 (3.3) | 5.2 (3.1)
  six weeks after operation at 30 ~ 40 degree | 11.6 (4.7) | 8.3 (5.1)
  six weeks after operation at 80 ~ 90 degree | 8.1 (2.8) | 5.8 (2.3)
  three months after operation at 10 ~ 20 degree | 4.9 (2.8) | 4.2 (2.7)
  three months after operation at 30 ~ 40 degree | 8.6 (5.0) | 7.4 (4.6)
  three months after operation at 80 ~ 90 degree | 6.3 (3.8) | 4.7 (3.1)
  six months after operation at 10 ~ 20 degree | 3.6 (3.4) | 3.8 (3.7)
  six months after operation at 30 ~ 40 degree | 11.4 (6.9) | 8.0 (4.0)
  six months after operation at 80 ~ 90 degree | 6.6 (4.5) | 5.5 (3.7)
Statistical Analysis 1: Comparison: MIS-TKA vs QS-TKA; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Secondary Outcome: HSS(Hospital for Special Surgery) Score of the Knee Joint
Description: Scale Name:score scale range:0~100,and a higher values represent a better outcome
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MIS-TKA | QS-TKA
Number analyzed (Participants) | 42 | 42
units on a scale
  one week after operation | 65.3 (9.1) | 68.4 (6.2)
  six weeks after operation | 69.6 (9.3) | 74.5 (7.7)
  three months after operation | 76.3 (9.3) | 77.8 (9.5)
  six months after operation | 81.1 (7.7) | 82.4 (5.8)
Statistical Analysis 1: Comparison: MIS-TKA vs QS-TKA; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

3. Secondary Outcome: VAS(Visual Analogue Scale/Score) of the Knee Joint
Description: Scale Name:score scale range:0~100,and a higher values represent a worse outcome
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MIS-TKA | QS-TKA
Number analyzed (Participants) | 42 | 42
units on a scale
  one week after operation | 2.5 (1.5) | 2.2 (1.7)
  six weeks after operation | 2.6 (1.8) | 2.7 (1.7)
  three months after operation | 1.8 (1.7) | 1.5 (1.2)
  six months after operation | 1.5 (1.0) | 1.4 (0.6)
Statistical Analysis 1: Comparison: MIS-TKA; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Six months
Description: Daily questionnaire, physical examination and laboratory for assessment.
Arm/Group | MIS-TKA | QS-TKA
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

LIMITATIONS AND CAVEATS:
Limitation was that the position reconstruction measurement mainly measures the difference of the reconstructed flex angle, while the reflex circuit and motion perception of the knee was not measured.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes